CLINICAL TRIAL: NCT05994261
Title: Evaluating Long-Term Feasibility of Cereset Research for Stressed Healthcare Workers
Brief Title: Cereset Research Long-Term Healthcare Worker Study
Acronym: LT-HW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Susanne Marcus Collins Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00099972
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Stress; Anxiety; Autonomic Dysregulation; Acoustic Stimulation; Hyperarousal; Health Personnel
Keywords: stress; anxiety; insomnia; Cereset Research; hyperarousal; brain electrical activity; autonomic dysregulation; neurotechnology; HIRREM; allostasis; neuromodulation; acoustic stimulation; COVID-19; healthcare worker
MeSH Terms: conditions — Anxiety Disorders; Primary Dysautonomias; Sleep Initiation and Maintenance Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study of long-term maintenance Cereset Research after an initial 4-session intervention bolus versus usual care control following an initial 4-session intervention bolus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cereset Research Tune-Up Intervention Group (Active Comparator): All study participants will receive 4 initial CR sessions. Afterwards, they will be randomized, and this group will receive an additional tune-up (maintenance) session every 6 weeks for one year. There will be a CR session at weeks 6, 12, 18, 24, 30, 36, 42, and 48.
  Interventions: Device: Cereset Research
- Cereset Research Control Group (Other): All study participants will receive 4 initial CR sessions. Afterwards, they will be randomized, and this group will continue their current care for 1 year with no additional CR sessions.
  Interventions: Device: Cereset Research

INTERVENTIONS:
Device: Cereset Research — The upgraded platform for medical research using the HIRREM technology has been rebranded as Cereset Research® (CR). This system uses the same core technology and algorithms to echo brainwaves in real-time using audible tones, as with HIRREM. The CR system also includes 64-bit processing architecture for faster feedback, the use of 4 sensors, and the use of standard protocols (with flexibility regarding the length and sequencing of the standard protocols), all done with eyes closed. Four sensors are applied to the scalp at a time. However, only two sensors are actively echoing feedback. The software automatically switches from one sensor pair to the other when needed. This reduces the number of sensor placement changes needed, resulting in shorter session time and fewer interruptions.

SUMMARY:
Randomized, controlled study of long-term maintenance Cereset Research after an initial 4-session intervention bolus versus usual care control following an initial 4-session intervention bolus.

DETAILED DESCRIPTION:
This randomized, controlled study will evaluate the effects of long-term Cereset Research maintenance intervention in healthcare workers with symptoms of stress in the post era of COVID-19. Healthcare workers of all types have been impacted personally, professionally, and financially by the pandemic and its aftermath, resulting in higher levels of stress and anxiety. Additional, brief, noninvasive, non-drug strategies are needed to help mitigate the effects of the acute trauma associated with the pandemic. The primary outcome will be change in Perceived Stress Scale (PSS) a measurement of how different situations affect feelings and perceived stress in the Intervention group compared to the Control Group. Data will also be collected on a variety of additional relevant symptoms including insomnia, anxiety and autonomic cardiovascular regulation, for which benefits have been shown in prior studies using High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM). Data collected will assess the long-term effects of a low dose Cereset Research (CR) approach (only 4 sessions) and the importance of long-term maintenance intervention versus control. The Intervention Group will then receive 1 session every 6 weeks beginning 6 weeks after the 4 session bolus is completed. The Control Group continues current care with no additional CR sessions. A successful outcome of reduced stress at 1 year in the Intervention Group vs. Control Group would suggest benefit for long-term maintenance intervention sessions. The effect of this approach on autonomic function and other self-reported symptoms will also be explored. This information will be useful for determining intervention schedules for direct clinical implementation of the intervention. The proposed study might also help to identify characteristics of individuals who may experience differential effects/benefits from application of CR and determine if intermittent "tune-up" sessions may prolong symptom improvement.

ELIGIBILITY:
Inclusion Criteria:

* Employed healthcare workers aged 18 years and older.
* Have availability and interest in participating in a 1 year study.
* Ability to comply with basic instructions and be able to sit still, comfortably during sessions.
* Experiencing symptoms of stress meeting threshold score on the Perceived Stress Scale (PSS ≥ 14).

Exclusion Criteria:

* No internet access, as some visits collected electronically
* Unable, unwilling, or incompetent to provide informed consent.
* Physically unable to come to the study visits, or to sit still, comfortably in a chair for up to 1 hour.
* Severe hearing impairment (because the subject will be using ear buds during CR).
* Weight is over the chair limit (400 pounds).
* Currently enrolled in another active intervention research study.
* Prior use of: HIRREM, HIRREM-SOP, Brainwave Optimization (BWO), Cereset, Cereset Research, Cereset Home, or a wearable configuration of the same (B2, or B2v2).
* Prior use of the following modalities within one month before enrollment: electroconvulsive therapy (ECT), prior use of transcranial magnetic stimulation (TMS), transcranial direct current stimulation (TDCS), alpha stimulation, eye movement desensitization and reprocessing (EMDR), brain spotting, neurofeedback, biofeedback, or deep brain stimulation (DBS).
* Known seizure disorder.
* Thoughts of active suicide within the last 3 months.
* Current medical student.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS) scores | Baseline to year 1
  The Perceived Stress Scale (PSS) is a ten-item psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale, with answers rated from 0-4, also includes a number of direct queries about current levels of experienced stress. Higher scores suggest increase perceived stress.

SECONDARY OUTCOMES:
Change in Insomnia Severity Index (ISI) scores | Baseline to year 1
  The severity of insomnia symptoms is measured using two self-report symptom inventories with each data collection visit. This includes the Insomnia Severity Index (ISI). The ISI is a 7-question measure, with responses from 0-4 for each question, yielding scores ranging from 0-28. The higher the score, the more suggestive of insomnia.
Change in Generalized Anxiety Disorder-7 (GAD-7) scores | Baseline to year 1
  The Generalized Anxiety Disorder-7 (GAD-7) is a seven-item screening tool for anxiety that is widely used in primary care. GAD-7 is a brief, reliable and valid measure of assessing generalized anxiety disorder. Higher scores suggest increased anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT05994261/ICF_000.pdf